CLINICAL TRIAL: NCT04104321
Title: A Phase 3, Multinational, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy PK, Kinetics and Safety of Aramchol in Nonalcoholic Steatohepatitis (NASH) With Open-Label Part
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Aramchol in Subjects With NASH (ARMOR)
Acronym: ARMOR
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis results from the open-label part of the study. The double blind portion of the study will be resumed once the study will continue.
Sponsor: Galmed Research and Development, Ltd. (Industry)
Responsible Party: Sponsor
Organization: Galmed Pharmaceuticals Ltd (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Aramchol-018
Record Dates: First submitted 2019-09-18; First posted 2019-09-26 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: fibrosis; liver fibrosis; diabetes; obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Liver Cirrhosis; Diabetes Mellitus; Obesity

STUDY DESIGN:
Intervention Model Description: In the Open Label part of the study, there will be a single group of 150 subjects (expected) all receiving Aramchol 300mg BID.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aramchol free acid (Experimental): Aramchol 300 mg oral tablet
  Interventions: Drug: Aramchol free acid
- Placebo (Placebo Comparator): Placebo matching oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aramchol free acid — Aramchol 300 mg BID
  Other Names: Two tablets of Aramchol free acid
  Arms: Aramchol free acid
Drug: Placebo — Placebo BID
  Other Names: Two tablet of Aramchol matching placebo
  Arms: Placebo

SUMMARY:
An Open-Label Part was added:

This part will enroll in selected sites which are less affected by the COVID-19 pandemic.

150 subjects with NASH and fibrosis confirmed by liver histology (F1-F3) will be randomized into 3 groups according to the post-baseline biopsy.

The objective of the Open-Label Part is:

* To evaluate the safety and PK of twice daily administration (BID) of Aramchol 300mg in subjects with NASH and liver fibrosis.
* To explore the kinetics of histological outcome measures and Non-Invasive Tests (NITs) associated with NASH and fibrosis for the treatment duration of 24, 48 and 72 weeks.

All patients will be allocated to Aramchol.

Double Blind Part:

This part is double blind, placebo controlled randomized in subjects with NASH and fibrosis stages 2-3 who are overweight or obese and have prediabetes or type 2 diabetes.

The primary objectives of this part of the study are to evaluate the effect of Aramchol as compared to placebo on NASH resolution, fibrosis improvement and clinical outcomes related to progression of liver disease.

Subjects will be randomized to receive Aramchol 300mg BID or matching placebo in a 2:1 randomization ratio.

This double-blind phase of the study will recruit patients once the study will be continued.

DETAILED DESCRIPTION:
A total of 150 subjects, including those already randomized to Aramchol 300 mg BID or Placebo, were to be randomized in a ratio of 1:1:1 to receive Aramchol 300 mg BID in the open-label (OL) part according to the grouping below:

Group A: The post-baseline liver biopsy was to be conducted at Week 24 Group B: The post-baseline liver biopsy was to be conducted at Week 48 Group C: The post-baseline liver biopsy was to be conducted at Week 72

In order to more comprehensively explore the kinetics of histological outcome measures (e.g., are there subjects who did not show improvement in outcome at Weeks 24, 48, or 72, but improved with longer duration of treatment), a second post-baseline liver biopsy sample was to be collected for subjects whose post-baseline liver biopsy at Weeks 24 or 48, or 72 did not show at least one stage improvement in fibrosis (fibrosis non-responders). The second post-baseline liver biopsy sample was to be collected one year later (i.e., at Weeks 72 or 96 or 120, respectively).

Subjects already randomized and ongoing in the PC part were given the option to switch to the OL part

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female age 18 to 75 years
2. Histological confirmation of NASH on a diagnostic liver biopsy by central reading of the slides (biopsy obtained within 6 months prior to randomization or during the screening period)
3. Total NAS Score 4 or more with at least 1 in each component of the NAS Score (steatosis ≥1 AND inflammation ≥1 AND ballooning ≥1)
4. Fibrosis Stage must be 2 or 3 (Open-Label Part may include up to 30 subjects with fibrosis stage 1)
5. Body mass index (BMI) between 25kg/m2 and 40 kg/m2 (Open Label part: BMI <40 kg/m2)
6. AST>20 IU/L
7. Type 2 diabetes mellitus or prediabetes (Open Label Part only: Type 2 diabetes or prediabetes is not an inclusion criteria)
8. For subjects with type 2 diabetes, glycemia must be controlled
9. Females of childbearing potential must practice a highly effective method of contraception throughout the study period and for 1 month after treatment discontinuation.
10. Able to understand the nature of the study and to provide signature of the written informed consent.

Key Exclusion Criteria:

1. Histologically documented liver cirrhosis (fibrosis stage 4)
2. Inability or unwillingness to undergo a liver biopsy
3. Abnormal synthetic liver function
4. ALT or AST >5× upper limit of normal (ULN)
5. Platelet count < 150,000mm3
6. Alkaline phosphatase ≥2× ULN
7. Known or suspected hepatocellular carcinoma (HCC)
8. Model for End-Stage Liver Disease (MELD) score > 12
9. Prior history or presence of decompensated liver disease
10. Other (acute or chronic) coexisting liver disease based on medical history and/or centralized review of liver histology)
11. Known alcohol and/or any other drug abuse or dependence in the last five years
12. Weight loss of more than 5% within 3 months prior to screening
13. History of bariatric surgery within 5 years of liver biopsy or planned surgery for weight reduction
14. Treatment with drugs that may cause NAFLD within 12 months prior to liver biopsy
15. Treatment with some anti-diabetic medications; Unless started prior to biopsy (timeframe depending on drug) and stable
16. Current or planned treatment with immunosuppressive drugs
17. Evidence of any other unstable or untreated clinically significant disease
18. Uncontrolled hypertension
19. Any other condition that in the opinion of the Investigator warrants exclusion from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2027-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yossi Gilgun-Sherki, PhD, MBA, Study Director — Executive Drug Development Consultant
Locations (2):
- United States (2):
  - The Public Health Trust of Miami-Dade County, Florida, dba the Jackson Health System, Miami, Florida
  - Texas Clinical Research Institute, LLC, Arlington, Texas

REFERENCES:
- [Result] Ratziu V, Yilmaz Y, Lazas D, Friedman SL, Lackner C, Behling C, Cummings OW, Chen L, Petitjean M, Gilgun-Sherki Y, Gorfine T, Kadosh S, Eyal E, Sanyal AJ. Aramchol improves hepatic fibrosis in metabolic dysfunction-associated steatohepatitis: Results of multimodality assessment using both conventional and digital pathology. Hepatology. 2025 Mar 1;81(3):932-946. doi: 10.1097/HEP.0000000000000980. Epub 2024 Jun 25. PMID 38916482

RESULTS

PARTICIPANT FLOW:
Groups:
- ARCON ITT: All subjects who were randomized to Aramchol
Period: Overall Study
Arm/Group | ARCON ITT
Started (157 subjects were randomized to receive Aramchol in either ARMOR Placebo part and/or the ARCON comprise the ARCON-Intent-To-Treat (ARCONITT) cohort) | 157
Subjects Randomized to the OL Part, Received Aramchol and Had Baseline and Post-baseline Biopsy (51 subjects had Baseline and post-baseline liver biopsy) | 51
Completed | 154 (Safety and tolerability were assessed based on all available data from 154 subjects according to their entire treatment duration in the study)
Not Completed | 3
Not completed — didn't take the study drug | 3

BASELINE CHARACTERISTICS:
Population: All patients who were randomized to Aramchol
Arm/Group | ARCON ITT
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 127
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 4
  White | 134
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 84
  Turkey | 25
  South Korea | 10
  Mexico | 7
  Chile | 6
  Spain | 5
  France | 5
  Canada | 5
  Australia | 4
  Belgium | 3
  Israel | 2
  United Kingdom | 1
Weight (kg) [Mean (Standard Deviation); unit: Kg] — Population: Data for 3 patients was missing
  Kg
    number analyzed (Participants) | 154
    (all) | 89 (15.2)
Body mass index (kg/m2) [Mean (Standard Deviation); unit: Kg/ M2] — Population: Height data was missing for 21 patients
  Kg/ M2
    number analyzed (Participants) | 136
    (all) | 32.7 (4.2)
Biopsy evaluation based on NASH CRN [Count of Participants; unit: Participants] — NASH Clinical Research Network (NASH CRN) is a scoring system developed and validated by a group of expert academic hepatopathologists. It comprises of 4 stages of fibrosis F0- No fibrosis, F1- mild fibrosis, F2- perisinusoidal fibrosis with portal/periportal fibrosis, F3- Bridging fibrosis and F4- Cirrhosis.
  Participants
    Baseline CRN fibrosis stage- F1 | 33
    Baseline CRN fibrosis stage- F2 | 34
    Baseline CRN fibrosis stage- F3 | 76
    Baseline CRN fibrosis stage- F4 | 8
    Not reported | 6
NAS score [Mean (Standard Deviation); unit: units on a scale] — Non alcoholic fatty liver disease (NAFLD) Activity Score (NAS) of the liver is a score that can range from 0 to 8 and is calculated by the sum of scores of steatosis (0-3), lobular inflammation (0-3) and hepatocyte ballooning (0-2).
  In patients with NAFLD, NAS score of ≥ 5 strongly correlated with a diagnosis of "definite non-alcoholic steatohepatitis (NASH)" whereas NAS ≤ 3 correlated with a diagnosis of "not NASH".
  units on a scale | 5.0 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Open Label Part: Improvement of Fibrosis Based on Liver Biopsy
Description: Improvement of fibrosis was defined by the following:
  1. One stage or more reduction in fibrosis stage as assesed by the NASH-CRN classification
  2. Ranked paired assessment between post-baseline compared to baseline biopsies (i,proved, worsened or stable fibrosis)
  3. Reduction in the the continous phenotypic Fibrosis composite severity (Ph-FCS) score ≥0.3 in absolute value or ≥25% in relative value
Time Frame: Up to 72 or 120 weeks
Population: 51 subjects performed a Baseline and post-baseline biopsy
Measure: Number (95% Confidence Interval); unit: percentage of participants improving
Groups:
- Aramchol: Aramchol 300 mg oral tablet
  Aramchol: Aramchol 300 mg BID
Arm/Group | Aramchol
Number analyzed (Participants) | 51
percentage of participants improving
  Fibrosis improvement NASH-CRN≥1 stage | 31.4 [19.1 to 45.9]
  NASH resolution without worsening of fibrosis | 26.5 [14.9 to 37.5]
  Fibrosis improvement by ranked assessment | 51.0 [36.6 to 65.2]
  Fibrosis improvement (absolute FCS score reduction ≥0.3 | 74.5 [60.4 to 85.7]
  Fibrosis improvement (relative FCS reduction by ≥25% AI cutoff) | 41.2 [27.6 to 55.8]

2. Primary Outcome: Double Blind Part: To Evaluate the Effect of Aramchol Compared to Placebo on Liver Histology by Assessing the Following Primary Endpoints. Study Was Suspended and Thus Results Are Expected 2027
Description: * Resolution of NASH defined as the Proportion (%) of subjects with resolution of NASH (defined by Ballooning of 0 and inflammation 0-1) and no worsening of liver fibrosis, or
  * Improvement in Fibrosis defined as the Proportion (%) of subjects with improvement in liver fibrosis greater than or equal to one stage and no worsening of steatohepatitis.
Time Frame: 72 weeks
Reporting Status: Not Posted, anticipated posting 2027-06

3. Primary Outcome: Double Blind Part: To Evaluate the Effect of Aramchol Compared to Placebo on Composite Long-term Outcome Study Was Suspended so Results Expected 2027
Description: Proportion (%) of subjects experiencing at least 1 of the following events: All-cause mortality, Liver transplant, Histological progression to cirrhosis, MELD score >15, Hospitalization due to hepatic decompensation event(s).
Time Frame: at End of Study, latest at 5 years from last subject's randomization
Reporting Status: Not Posted, anticipated posting 2027-06

ADVERSE EVENTS:
Time Frame: Up to 124 weeks
Groups:
- Patients Randomized to the OL Part of the ARMOR Study: Patients that have been randomized to the OL part of the ARMOR study and receiving Aramchol 300 mg BID
Arm/Group | Patients Randomized to the OL Part of the ARMOR Study
All-Cause Mortality (participants affected / at risk) | 154/154
Serious Adverse Events (participants affected / at risk) | 1/154
Other Adverse Events (participants affected / at risk) | 27/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Randomized to the OL Part of the ARMOR Study (N=154)
coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Post-procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Post-procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Lung adenocarcinoma was diagnosed in a subject with a known lung nodule
Dizziness (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pulmonary fibrosis exacerbation occurred in a subject with idiopathic pulmonary fibrosis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Randomized to the OL Part of the ARMOR Study (N=154)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10)
COVID-19 (Infections and infestations) | 27 (29)
Constipation (Gastrointestinal disorders) | 8 (10)
Headache (Nervous system disorders) | 12 (18)
Hypertension (Cardiac disorders) | 10 (10)
Nausea (Gastrointestinal disorders) | 8 (8)
Procedural pain (Surgical and medical procedures) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT04104321/Prot_SAP_000.pdf